CLINICAL TRIAL: NCT06902285
Title: Use of Magnesium-L-Threonate to Improve Subjective Sleep Quality After Total Joint Arthroplasties: Randomized Controlled Clinical Trial
Brief Title: Magnesium-L-Threonate for Sleep Quality Post-Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20240578
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Sleep; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — threonic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium L Threonate Group (Experimental): Participants in this group will receive the Magnesium L Threonate intervention for up to 6 weeks postoperatively
  Interventions: Drug: Magnesium Threonate
- Control Group (Placebo Comparator): Participants in this group will receive the placebo comparator for up to 6 weeks postoperatively
  Interventions: Other: Control

INTERVENTIONS:
Drug: Magnesium Threonate — Participants will receive a daily 145 mg pill by mouth 30 minutes before going to sleep
  Arms: Magnesium L Threonate Group
Other: Control — Participants will receive two sugar pills daily by mouth 30 minutes before going to sleep
  Arms: Control Group

SUMMARY:
The study team is conducting a study to see if Magnesium-L-Threonate (MgT) can help improve how well participants sleep and reduce pain after total joint replacement surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total knee or hip arthroplasty at the University of Miami Hospital
* Patients > 18 years of age
* Subjects must be capable of providing informed consent
* English or Spanish-speaking

Exclusion Criteria:

* Previous total joint arthroplasty at the surgical site
* History of sleeping disorders, including narcolepsy, sleep apnea, insomnia, parasomnias, and restless leg syndrome.
* History of Complex Regional Pain Syndrome in ipsilateral extremity
* History of demyelinating disorder or neurologic deficit in the affected extremity
* History of psychiatric disorders that could impact sleep, such as untreated depression, bipolar disorder, or schizophrenia.
* Participants taking medications known to cause significant sedation or insomnia.
* Pregnant or breastfeeding
* Being treated for a diagnosis other than primary osteoarthritis (e.g. pelvic/femur fracture)
* Patients with known substance use disorder within 6 months of surgery
* Liver Failure, via clinical diagnosis or international normalized ratio greater than 1.5 or Prothrombin time greater than 40
* Chronic Kidney Disease or glomerular filtration rate less than 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Epsworth Sleepiness Score | 2 weeks, 4 weeks, 6 weeks
  Score ranging from 0-24 with higher scores indicating greater sleepiness.
Change in Pittsburgh Sleep Quality Index (PSQI) | 2 weeks, 4 weeks, 6 weeks
  The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep

SECONDARY OUTCOMES:
Change in Morphine Milligram Equivalent Prescribed | 2 weeks, 4 weeks, 6 weeks
  Measured in milligram equivalents
Patient-reported outcome measured by Knee Injury and Osteoarthritis Outcome Score | 6 weeks
  The total score ranges from 0-100. Lowers scores indicate a healthier knee
Medication Compliance measured in number of days study medication taken | 6 weeks
  Medication compliance as measured by number of days taking study medication

CONTACTS AND LOCATIONS:
Overall Officials: Victor H Hernandez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No